CLINICAL TRIAL: NCT01040312
Title: A Prospective Observational Study of the Efficacy and Safety of CPT-11 Plus Platinum Analogues Regimens for UGT1A1 Genotype Guided Patients With Several Solid Tumors
Brief Title: An Observational Study of CPT-11 Plus Platinum Analogues Regimens and UGT1A1 Genotypes in Solid Tumors
Status: Completed | Type: Observational
Sponsor: Daiichi Sankyo Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Daiichi Sankyo (Industry)
Other Study IDs: TOP009-062; 090946 (Other: JAPIC ID)
Record Dates: First submitted 2009-12-23; First posted 2009-12-29 (Estimated); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Small Cell Lung Cancer; Non-small Cell Lung Cancer; Cervical Cancer; Ovarian Cancer; Gastric Cancer (Inoperable and Recurrent)
Keywords: UGT1A1, irinotecan
MeSH Terms: conditions — Small Cell Lung Carcinoma; Carcinoma, Non-Small-Cell Lung; Uterine Cervical Neoplasms; Ovarian Neoplasms; Stomach Neoplasms; Recurrence | interventions — Irinotecan; Cisplatin; Carboplatin; nedaplatin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — white cells
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- UGT1A1 genotyped patients: UGT1A1 genotyped patients receive CPT-11 with platinum analogues
  Interventions: Drug: CPT-11; Drug: Platinum analogues

INTERVENTIONS:
Drug: CPT-11 — CPT-11 blocks certain enzymes needed for cell division and DNA repair, and it may kill cancer cells. It is a type of topoisomerase inhibitor and a type of camptothecin analog.
  Other Names: Camptosar; Topotecin
Drug: Platinum analogues — Platinum compounds produce changes in DNA structure, which causes cancer cell death (apoptosis). They are typically used alone or in combination with other chemotherapy drugs.
  Other Names: Cisplatin; Carboplatin; Nedaplatin

SUMMARY:
The purpose of this study is to examine the correlation between UGT1A1 genotypes and the safety of CPT-11 plus platinum analogues (cisplatin, carboplatin and nedaplatin) regimens for patients with lung cancer, cervical cancer, ovarian cancer and gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* Has small cell lung cancer, non-small cell lung cancer, cervical cancer, ovarian cancer and/or gastric cancer
* Has UGT1A1 genotype *1/*6, *1/*28, *6/*6, *28/*28 and *6/*28
* Is receiving CPT-11 plus platinum analogue (cisplatin, carboplatin and nedaplatin) regimens (with or without molecular targeted agents)

Exclusion Criteria:

* Has contraindication for CPT-11
* Has an Eastern Cooperative Oncology Group (ECOG) performance score (PS) of 3-4

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients in Japan with small cell lung cancer, non-small cell lung cancer, cervical cancer, ovarian cancer and/or gastric cancer treated with CPT-11 plus platinum analogues (cisplatin, carboplatin and nedaplatin) in clinical practice
Sampling Method: Probability Sample
Enrollment: 321 (Actual)
Dates: Start 2009-10-15 (Actual); Primary Completion 2014-09-29 (Actual); Study Completion 2015-09-02 (Actual)

PRIMARY OUTCOMES:
Number of Participants with UGT1A1 Genotype with Severe Toxicities Induced by CPT-11 with Platinum Analogues | within 6 months

SECONDARY OUTCOMES:
Response Rate of Participants with UGT1A1 genotype to CPT-11 with Platinum Analogues | within 6 months
Duration of Response to CPT-11 with Platinum Analogues in Participants with UGT1A1 Genotype | within 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Study Leader, Study Director — Daiichi Sankyo
Locations (1):
- Department of Obstetrics and Gynecology, National Defense Medical College Hospital, Tokorozawa, Japan

IPD SHARING:
Plan to Share IPD: No